CLINICAL TRIAL: NCT02993887
Title: The Effects of Resourcefulness Training Intervention and Decentering on Self-Management of Stress in Caregivers of Children With Complex Chronic Conditions Dependent on Lifesaving Medical Technology: A Pilot Study
Brief Title: Resourcefulness Training and Decentering on Self-Management in Caregivers of Technology Dependent Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Valerie Toly, Assistant Professor of Nursing, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10-16-10
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Caregiver; Mindfulness; Mechanical Ventilation Pressure High; Gastrostomy; Chronic Illness
Keywords: Caregiver; Technology Dependent Children; Resourcefulness; Mindfulness
MeSH Terms: conditions — Chronic Disease | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Placebo Comparator): Mindfulness (Decentering) only using the Stop, Breathe, Think Smart Phone application
  Interventions: Behavioral: Mindfulness
- Resourcefulness and Mindfulness (Experimental): Resourcefulness Training (a cognitive behavioral intervention that teaches self-help and help-seeking skills) and Mindfulness using the Stop, Think, Breathe app.
  Interventions: Behavioral: Resourcefulness Training; Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Resourcefulness Training — This intervention will include a one time face to face instruction on Resourcefulness Training that entails 8 self-help and help-seeking skills plus viewing short video vignettes of caregivers describing application of the resourcefulness skills. In addition, participants will use daily journaling to describe application of the resourcefulness skills in their daily caregiving with their technology-dependent child.
  Arms: Resourcefulness and Mindfulness
Behavioral: Mindfulness — The mindfulness intervention will include the use of an app daily via Stop, Think, Breathe.

SUMMARY:
The investigators will conduct a randomized clinical trial pilot study to examine the effectiveness of a theoretically based intervention (called ReMind) encompassing two key components: (a) Resourcefulness Training for parent caregivers, and (b) daily mindfulness meditation delivered using a smart phone application (Stop, Breathe & Think™) with an intervention (Mind Only) that consists only of daily mindfulness meditation. Both components of the intervention have been tested separately (but not combined) and both interventions can be self-tailored, which meets the vital need for these caregivers to engage in self-management activities when it is convenient for them. The investigators will test the two arms of the intervention in 30 parents of technology-dependent children, 15 parents in each group. The investigators will collect mixed data at baseline, 3 months and 6 months after subject enrollment to describe changes in proximal and distal outcomes. The investigators aim to:

1. Evaluate the intermediate (3 month) and long-term (6 month) effects of the ReMind and Mind Only interventions on study mediators (HPA Axis Function and stress, cognitive factors, resourcefulness) and determine if there are different effects between ReMind and Mind Only interventions.
2. Evaluate the differences in distal psychological (Mental Health Related Quality of Life, Depressive Cognitions, Depressive Symptoms, Anxiety, Caregiver Burden), physical (Physical Health Related Quality of Life), and cost outcomes between subjects in the ReMind and Mind Only arms over time.
3. Determine the moderating effects of parents' social support, demographics (age, gender, family income) and children's functional status on (a) proximal outcomes and the relationship between (a) the intervention arm and distal outcomes, and (b) HPA Axis Function, stress, cognitive factors and distal outcomes.
4. Evaluate the impact of decentering on the association between the interventions and the proximal and distal outcomes.
5. Explore differences in neurological processing (DMN and TPN) and decentering in proximal and distal outcomes associated with each intervention.

DETAILED DESCRIPTION:
Design Overview. The investigators will conduct a two-arm Randomized Clinical Trial to compare the effects of the ReMind with the Mind interventions on psychological and physical health outcomes and cognitive task switching between the DMN and TPN neural networks in Functional Magnetic Resonance Imaging (fMRI) and Diffusion Tensor Imaging (DTI). The full ReMind intervention involves daily self-tailored mindful meditation application focused on kindness and compassion for 4 weeks with self-selected frequency of use thereafter. The application that is being used is theoretically constructed and tested and can be delivered on a smart phone app for free (iPad, computer as well). ReMind also includes five resourcefulness training aspects: 1) one face-to-face session for teaching social (help-seeking) and personal (self-help) resourcefulness skills, 2) ongoing web access to video vignettes of parents of technology-dependent children describing the application of resourcefulness skills in daily life, 3) 4 weeks of skills' reinforcement using daily journal writing by the parents, 4) weekly phone calls from the intervention nurse over 4 weeks after face-to-face intervention training. The Mind Only intervention includes only the meditation component. Thus, the investigators will be able to see if the addition of Resourcefulness Training will significantly impact proximal outcomes (self management behaviors) such as appraised sleep quality, positive health practices and distal outcomes such as psychological health (Mental Health Related Quality of Life, depressive cognitions, anxiety, caregiver burden), physical health (Physical Health Related Quality of Life), and economic costs.

Sample. A purposive sample of 30 parent caregivers of technology-dependent children (n=15 ReMind, n=15 Mind Only) seen at outpatient clinics (Pulmonology, Gastroenterology, Trach/Vent). The investigators have used this patient population in prior work. Given the availability of potential subjects and the investigator's experience with this population, the investigators anticipate little difficulty in recruiting 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. parent (biological, adoptive, or foster mother, father, grandmother, or grandfather) caregiver for a child aged ≤17 years dependent on medical technology (mechanical ventilators, intravenous nutrition/medication, respiratory or nutritional support) at home;
2. aged ≥18 years;
3. able to speak and understand English.

   Exclusion Criteria:

   1. currently practicing mindfulness-based interventions (yoga, meditation, deep breathing)

   2 history of a medical condition or procedure that is contraindicated for imaging (i.e. cardiac pacemaker, sternal wires, or metal implants);

   3 claustrophobia requiring anxiolytics or sedation

   4 Pregnancy at time of recruitment.

   5 If participant becomes pregnant during the follow up period the participant will be excluded from all imaging studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Mental & Physical Health Related Quality of Life at 3 Months & 6 Months | Measured at baseline with follow up at 3 months, 6 months
  Measure using the Patient Reported Outcomes Measurement Information System (PROMIS)-29

SECONDARY OUTCOMES:
Change from Baseline Appraised Sleep Quality at 3 months and 6 months | Measured at baseline with follow up at 3 months, 6 months
  Measure using Pittsburgh Sleep Quality Index
Change from Baseline Positive Health Practices at 3 months and 6 months | Measured at baseline with follow up at 3 months, 6 months
  Measure using Personal Lifestyle Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Valerie A Toly, PhD, Principal Investigator — Case Western Reserve University, Frances Payne Bolton School of Nursing
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moore SM, Musil CM, Alder ML, Pignatiello G, Higgins P, Webel A, Wright KD. Building a Research Data Repository for Chronic Condition Self-Management Using Harmonized Data. Nurs Res. 2020 Jul/Aug;69(4):254-263. doi: 10.1097/NNR.0000000000000435. PMID 32205788